CLINICAL TRIAL: NCT06681714
Title: Kalp Yetersizliği Somatik Algı Ölçeğinin Türkçe Geçerlik Ve Güvenirlik Çalışması
Brief Title: The Validity and Reliability of the Turkish Version of the Heart Failure Somatic Perception Scale
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Hacettepe University
Other Study IDs: SBA 24/702
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart Failure: Patients with heart failure

SUMMARY:
The aim of this study is to evaluate The Validity and Reliability of the Turkish Version of the Heart Failure Somatic Perception Scale in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure is a global health issue that serves as the endpoint for many cardiovascular conditions, particularly coronary heart disease and hypertension. Common symptoms of heart failure include fatigue, dyspnea, edema, cough, lack of energy, orthopnea, paroxysmal nocturnal dyspnea, palpitations, and dizziness. These symptoms significantly affect the health-related quality of life of individuals with heart failure, especially in the palliative phase of the disease. Additionally, heart failure patients often experience physical limitations, reduced quality of life, and an increased rate of hospital admissions due to symptoms such as breathlessness and fatigue. The Heart Failure Somatic Perception Scale assesses the presence and severity of 18 common physical signs and symptoms of heart failure (e.g. chest pain), as well as dyspnea and its impact on daily activities through six items. Robust and rigorous measures are needed to assess the complexity of heart failure symptoms, and evidence suggests that evaluating a broad range of heart failure symptoms can be beneficial in guiding rehabilitation approaches, clinical decision-making, and survival prediction.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of heart failure. Use of optimal pharmacological treatment according to current guidelines for at least 3 months.

Functional capacity classified as New York Heart Association (NYHA) Class I-IV (ambulatory).

Age 18 or older. Ability to cooperate with measurements.

Exclusion Criteria:

Known cognitive impairment. Having undergone acute coronary syndrome, percutaneous coronary intervention, or heart surgery within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-06-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
The Heart Failure Somatic Perception Scale | 1 day
  The Heart Failure Somatic Perception Scale comprises 18 items that assess how much the main signs and symptoms of heart failure have distressed the individual over the past week.
  Each item is rated on a five-point Likert scale, ranging from 0, indicating "did not experience this symptom," to 5, indicating "severe distress." The total score is obtained by summing the scores of all items, yielding a range from 0 to 90.
  A higher score indicates a greater impact of heart failure symptoms on the patient's life.
  Turkish version of The Heart Failure Somatic Perception Scale will be applied.

SECONDARY OUTCOMES:
The Heart Failure Symptom Status Scale | 1 day
  The Heart Failure Symptom Status Scale is designed to assess the presence, frequency, severity, and impact of the seven most common symptoms in patients with heart failure.
  Patients evaluate the presence, frequency, and severity of symptoms such as dyspnea, orthopnea, fatigue, chest pain, edema, sleep disturbances, dizziness, or lightheadedness using a four-point Likert scale.
  The total score attainable on this scale ranges from 0 to 84.
Mini mental test | 1 day
  The Mini-Mental test was developed to assess cognitive impairment in adults. It is structured under five main categories: orientation, registration memory, attention and calculation, recall, and language. The test is scored on a total of 30 points. Individuals scoring 17 or below are classified as having severe dementia, those scoring between 18 and 23 are classified with mild dementia, and individuals scoring between 24 and 30 are considered not to have dementia.
The MacNew Heart Disease-Specific Quality of Life Questionnaire | 1 day
  The MacNew Heart Disease-Specific Quality of Life Questionnaire is an internationally recognized tool for measuring health-related quality of life in patients with Coronary Artery Disease (CAD).
  The questionnaire is designed to assess how physical, emotional, and social functions, as well as daily activities, are affected by CAD. The questionnaire consists of three subscales: physical limitation, emotional function, and social function, with a total of 27 items. Subscale scores are calculated by averaging the responses to the relevant items. For each subscale and for the total score, the lowest possible score is 1 and the highest is 7, with higher scores indicating better quality of life.
Charlson Comorbity Index | 1 day
  It is a mortality scoring system that includes 19 comorbidity diagnostic groups. This index is frequently used as an assessment tool for evaluating comorbidities. A score of "1 point" is assigned for the presence of myocardial infarction, congestive heart failure, peripheral vascular diseases, cerebrovascular disease, dementia, chronic pulmonary disease, connective tissue disease, ulcer disease, mild liver disease, and diabetes. A score of "2 points" is given for conditions such as hemiplegia, moderate/severe renal disease, diabetes with end-organ damage, tumors, leukemia, and malignant lymphoma. A score of "3 points" is assigned for moderate/severe liver disease, and "6 points" is given for the presence of metastatic solid tumors and AIDS. The total score is calculated by summing the individual scores, with higher scores indicating more serious conditions and a worse prognosis.
The Minnesota Living with Heart Failure Questionnaire | 1 day
  The Minnesota Living with Heart Failure Questionnaire consists of 21 items that examine the physical and emotional dimensions of heart failure. Items 2, 3, 4, 5, 6, 7, 12, and 13 assess the physical dimension, while items 17, 18, 19, 20, and 21 assess the emotional dimension. Each item is scored on a scale from 0 to 5, with a maximum possible score of 105. Higher scores indicate poorer quality of life.
The Fatigue Severity Scale | 1 day
  The Fatigue Severity Scale is a questionnaire designed to measure the severity of fatigue over the past week. It consists of 9 items, each rated on a scale from 0 to 7. The total score is obtained by summing the responses to all items and dividing the sum by 9. A score of 4 or higher typically indicates severe fatigue.
The Leicester Questionnaire | 1 day
  The Leicester Cough Questionnaire is a health-related quality of life tool specifically designed for chronic cough. It is a self-administered, easy-to-use form that evaluates the impact of chronic cough on physical, psychological, and social aspects of life. The questionnaire consists of 19 items across these three domains, and it uses a 7-point Likert scale for responses.
  Higher scores on the LCQ indicate that the individual is less affected by the cough, reflecting better overall health. The total score is the sum of the scores from the physical, psychological, and social domains.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PT, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)